CLINICAL TRIAL: NCT06722079
Title: A Comparative Study of the Therapeutic Effect of PEGylated Recombinant Human Growth Hormone(PEG-rhGH) Injection on Turner Syndrome in a Clinical Trial and Short-acting Recombinant Human Growth Hormone in a Real World Study
Brief Title: A Real-world Study of Long-acting Growth Hormone Injection for Turner Syndrome
Status: Completed | Type: Observational
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Tongji Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Gensci032-401
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PEG-rhGH injection: The group of Turner syndrome patients treated with a dose of 0.2 mg/kg/ week in GenSci032-02 clinical trial.
- rhGH injection: Part A control group: a group of Turner syndrome patients treated with rhGH who met the inclusion criteria of the RWS study population from participating research centers in China.
  Part B control group: studies of rhGH treatment for Turner syndrome performed abroad that met all MA inclusion criteria and did not meet any MA exclusion criteria.

SUMMARY:
This study is divided into two parts:

Part A: A multicenter, retrospective, observational study to evaluate the effectiveness of PEG-rhGH in the treatment of Turner syndrome with domestic real-world data on rhGH as external controls. The collection and arrangement of real world data is the content of the real world study (RWS); Part B: Meta analysis (MA) was conducted based on the previous literatures on rhGH in the treatment of Turner syndrome, and MA results were used as external controls to evaluate the effectiveness of PEG-rhGH.

Real-world data on rhGH treatment of Turner syndrome in China were obtained from the HIS system and/or paper medical records of participating domestic centers and/or photocopied/printed medical records of other hospitals. Data on the efficacy of PEG-rhGH injection in the treatment of Turner syndrome were obtained from the 0.2mg /kg/ week group in the Phase II clinical trial of PEG-rhGH injection in the treatment of Turner syndrome (multicenter, randomized, blank control, superior efficacy) conducted by Changchun GeneScience Pharmaceutical Co., Ltd (Protocol number: GenSci032-02, version date: April 27, 2015). The MA study data of rhGH in the treatment of Turner syndrome in foreign countries came from the relevant literature retrieved from the approved drug database of FDA, PubMed and Web of Science database.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Turner syndrome by a clinician;
* The first treatment was short-acting rhGH, and the first administration date was not earlier than July 1, 2008;
* Follow-up data are available at the center before the first dosing and after at least one dosing.

Exclusion Criteria:

● None.

Ages: 0 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — The indication in this study is Turner syndrome, which only occurred in females.
Study Population: The indication in this study is Turner syndrome, which only occurred in females.
Sampling Method: Non-Probability Sample
Enrollment: 743 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Change in height standard deviation scores (HT SDS) after 1 year (52 weeks) of treatment compared to before (i.e., baseline) (ΔHT SDS). | Week 52
  Change in height standard deviation scores (HT SDS) after 1 year (52 weeks) of treatment compared to before (i.e., baseline) (ΔHT SDS).

SECONDARY OUTCOMES:
The annualized height velocity (AHV, cm/ year) after 1 year (52 weeks) of treatment. | Week 52
  The annualized height velocity (AHV, cm/ year) after 1 year (52 weeks) of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: xiaoping Luo, Doctor, Study Chair — Tongji hospital affiliated to tongji medicalcollege of huazhong university of science＆technology
Locations (1):
- Tongji hospital affiliated to tongji medicalcollege of huazhong university of science＆technology, Wuhan, Hubei, China